CLINICAL TRIAL: NCT00365729
Title: Evaluation of Viral Load Determination and Other Biomarkers of High Risk HPV-Types as a Marker for Progression of Perianal HPV-infections in HIV-positive Men Who Have Sex With Men
Brief Title: Viral Load Determination and Biomarkers of High Risk Human Papillomavirus (HPV) - Types in HIV-positive Men
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Deutsche Luft und Raumfahrt (Other Government)
Responsible Party: Principal Investigator, Alexander Kreuter, Prof. Dr., Deutsche Luft und Raumfahrt
Other Study IDs: 01 KI 0211
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: HIV Infections; Papillomavirus Infections; Anal Intraepithelial Neoplasia
Keywords: genitoanal HPV infection; HIV infection
MeSH Terms: conditions — HIV Infections; Papillomavirus Infections | interventions — Viral Load

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Anogenital smears

INTERVENTIONS:
Behavioral: Smear and biopsy testing for HPV-types and viral load — Smear and biopsy testing for HPV-types and viral load

SUMMARY:
Human papillomavirus (HPV)-infection belongs to the most common sexually transmitted diseases worldwide. HIV-infected men having sex with men (MSM) are strongly associated with a higher prevalence of genital HPV-infection, a higher incidence of anal intraepithelial neoplasia (AIN), and, consecutively, an increased risk for anal cancer. Since the introduction of highly active antiretroviral therapy (HAART), the incidence of several viral-associated neoplasias has significantly fallen in HIV-infected individuals. At the beginning of the era of HAART, a justified hope existed that genitoanal HPV-related neoplasias would also decrease based on the success of HAART-induced immune restoration. However, HAART seems to have only a small impact on the natural history of AIN as observed in a cohort of HIV-positive MSM before and after the initiation of HAART.

As AIN and cancer precursor lesions of the cervix, cervical intraepithelial neoplasia, share distinct clinical similarities, cytologic smear testing for AIN has been recommended to detect and treat early lesions. Thus, this prospective study mainly focuses on the predictive value of HPV-DNA load for the development and clinical progression of AIN in HIV-infected MSM. Moreover, the course of HPV viral load under therapy for anal intraepithelial neoplasia, e.g. topical treatment with imiquimod, will be evaluated. Additionally, immunohistochemical determination of several proliferative biomarkers, as well as cytokines, will be performed.

DETAILED DESCRIPTION:
Compared to the general population the incidence of anal intraepithelial neoplasia (AIN) and anal carcinoma (AC) amongst men who have sex with men (MSM) is extremely high (above 70/100,000). While many opportunistic infections have declined since the introduction of highly active antiretroviral therapy (HAART), the incidence of AC has not fallen. In contrast, the HAART-related improvement of survival seems to result in an increased risk of AC in HIV-infected MSM. Screening for cervical intraepithelial neoplasia (CIN) with cervical cytology and early treatment has resulted in a significant decline in the incidence of cervical carcinoma. Like cervical cancer, AC may be preventable through identification and treatment of its precursors. Nevertheless, there has never been an effort to implement an anal cytology screening program for HIV-infected MSM. Persistent cervical infection with high-risk HPV-types is indicative for the development of CIN and cervical cancer. As the prevalence of genital HPV-infections in HIV-infected women and men is very high (up to > 90%), the predictive value of qualitative HPV-DNA detection is limited for cervical cancer or AC prevention. However, several studies have shown that the number of HPV-DNA copies in cervical scrapes may be predictive of the severity of underlying cervical dysplasia. Thus, this prospective study mainly focuses on the predictive value of HPV-DNA load for the development and clinical progression of AIN in HIV-infected MSM. Besides, HPV-E6/E7-oncogen-expression using RT-polymerase chain reaction (RT-PCR) will be determined. Moreover, the course of HPV viral load under therapy for anal intraepithelial neoplasia, e.g. topical treatment with imiquimod, will be evaluated. Additionally, immunohistochemical determination of several proliferative biomarkers as well as cytokines will be performed.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected patients

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: HIV-positive men who have sex with men
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2003-10; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Spectrum of HPV types, HPV viral loads, and associated clinical lesions | swabs will be obtained approximately every 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Norbert H Brockmeyer, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum; Alexander Kreuter, MD, Principal Investigator — Department of Dermatology, Ruhr University Bochum
Locations (2):
- Germany (2):
  - Department of Dermatology, Ruhr University Bochum, Bochum, North Rhine-Westphalia
  - Institute of Virology, Cologne, North Rhine-Westphalia

REFERENCES:
- [Background] Kreuter A, Reimann G, Esser S, Rasokat H, Hartmann M, Swoboda J, Conant MA, Tschachler E, Arasteh K, Altmeyer P, Brockmeyer NH. [Screening and therapy of anal intraepithelial neoplasia (AIN) and anal carcinoma in patients with HIV-infection]. Dtsch Med Wochenschr. 2003 Sep 19;128(38):1957-62. doi: 10.1055/s-2003-42360. German. PMID 14502448
- [Result] Kreuter A, Brockmeyer NH, Hochdorfer B, Weissenborn SJ, Stucker M, Swoboda J, Altmeyer P, Pfister H, Wieland U. Clinical spectrum and virologic characteristics of anal intraepithelial neoplasia in HIV infection. J Am Acad Dermatol. 2005 Apr;52(4):603-8. doi: 10.1016/j.jaad.2004.11.026. PMID 15793509
- [Result] Kreuter A, Hochdorfer B, Stucker M, Altmeyer P, Weiland U, Conant MA, Brockmeyer NH. Treatment of anal intraepithelial neoplasia in patients with acquired HIV with imiquimod 5% cream. J Am Acad Dermatol. 2004 Jun;50(6):980-1. doi: 10.1016/j.jaad.2003.12.025. No abstract available. PMID 15153912
- [Result] Kreuter A, Brockmeyer NH, Weissenborn SJ, Wafaisade A, Pfister H, Altmeyer P, Wieland U; German Competence Network HIV/AIDS. 5% imiquimod suppositories decrease the DNA load of intra-anal HPV types 6 and 11 in HIV-infected men after surgical ablation of condylomata acuminata. Arch Dermatol. 2006 Feb;142(2):243-4. doi: 10.1001/archderm.142.2.243. No abstract available. PMID 16490857
- [Result] Kreuter A, Wieland U, Brockmeyer N. [Anal carcinoma and anal intraepithelial neoplasia in HIV-infections]. J Dtsch Dermatol Ges. 2006 Jul;4(7):611-2. doi: 10.1111/j.1610-0387.2006.06766.x. No abstract available. German. PMID 16883662
- [Result] Kreuter A, Brockmeyer NH, Pfister H, Altmeyer P, Wieland U; Competence Network HIV/AIDS. Human papillomavirus type 26-associated periungual squamous cell carcinoma in situ in a HIV-infected patient with concomitant penile and anal intraepithelial neoplasia. J Am Acad Dermatol. 2005 Oct;53(4):737-9. doi: 10.1016/j.jaad.2005.03.022. No abstract available. PMID 16198810
- [Derived] Kreuter A, Potthoff A, Brockmeyer NH, Gambichler T, Swoboda J, Stucker M, Schmitt M, Pfister H, Wieland U; German Competence Network HIV/AIDS. Anal carcinoma in human immunodeficiency virus-positive men: results of a prospective study from Germany. Br J Dermatol. 2010 Jun;162(6):1269-77. doi: 10.1111/j.1365-2133.2010.09712.x. Epub 2010 Feb 22. PMID 20184584
- [Derived] Kreuter A, Brockmeyer NH, Weissenborn SJ, Gambichler T, Stucker M, Altmeyer P, Pfister H, Wieland U; German Competence Network HIV/AIDS. Penile intraepithelial neoplasia is frequent in HIV-positive men with anal dysplasia. J Invest Dermatol. 2008 Sep;128(9):2316-24. doi: 10.1038/jid.2008.72. Epub 2008 Apr 3. PMID 18385760
- [Derived] Kreuter A, Wieland U, Gambichler T, Altmeyer P, Pfister H, Tenner-Racz K, Racz P, Potthoff A, Brockmeyer NH; German Network of Competence HIV/AIDS. p16ink4a expression decreases during imiquimod treatment of anal intraepithelial neoplasia in human immunodeficiency virus-infected men and correlates with the decline of lesional high-risk human papillomavirus DNA load. Br J Dermatol. 2007 Sep;157(3):523-30. doi: 10.1111/j.1365-2133.2007.08004.x. Epub 2007 Jun 15. PMID 17573882
- [Derived] Wieland U, Brockmeyer NH, Weissenborn SJ, Hochdorfer B, Stucker M, Swoboda J, Altmeyer P, Pfister H, Kreuter A. Imiquimod treatment of anal intraepithelial neoplasia in HIV-positive men. Arch Dermatol. 2006 Nov;142(11):1438-44. doi: 10.1001/archderm.142.11.1438. PMID 17116834